CLINICAL TRIAL: NCT02031913
Title: Association Between Insulin Resistance and Hepatic Fibrosis in Combined Chronic Hepatitis B and Non-alcoholic Fatty Liver Disease
Brief Title: Prospective Cohort Study of Association of Insulin Resistance/Steatosis With Hepatic Fibrosis in CHB and NAFLD
Status: Completed | Type: Observational
Sponsor: Seoul National University Boramae Hospital (Other)
Responsible Party: Principal Investigator, Won Kim, M.D, PhD, Seoul National University Boramae Hospital
Other Study IDs: HBV_FL
Record Dates: First submitted 2014-01-08; First posted 2014-01-09 (Estimated); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Chronic Hepatitis B; Hepatic Fibrosis; Fatty Liver
Keywords: Chronic hepatitis B; Hepatic fibrosis; Steatosis
MeSH Terms: conditions — Hepatitis B, Chronic; Liver Cirrhosis; Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples Without DNA — We intended to collect sera from registered subjects, but no biospecimens are to be retained yet.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HBV without FL: Chronic hepatitis B without steatosis
- HBV with FL: Chronic hepatitis B patients with steatosis

SUMMARY:
Hepatic steatosis and insulin resistance are associated with severity of fibrosis in non-alcoholic fatty liver disease (NAFLD) and chronic hepatitis C. However, clinical significance of steatosis and insulin resistance on fibrosis in chronic hepatitis B (CHB) is not well established. The aim was to investigate the relationship between insulin resistance, hepatic steatosis, and fibrosis in patients with CHB.

DETAILED DESCRIPTION:
acoustic radiation force impulse elastography

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B patients
* With evidences of hepatic steatosis on ultrasonography or pathology

Exclusion Criteria:

* significant alcohol consumption or other known liver diseases

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic hepatitis B patients who showed evidences of hepatic steatosis on ultrasonography
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2013-01; Primary Completion 2022-11 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Insulin resistance and fibrosis indices | one year
  Measurement for insulin resistance and fibrosis index for hepatic fibrosis assessment

CONTACTS AND LOCATIONS:
Overall Officials: Won Kim, Professor, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Seoul Metropolitan Government Seoul National University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No